CLINICAL TRIAL: NCT06669689
Title: The Impact of Anesthesia and Positioning on Cerebral Blood Flow and Pressure in Patients Undergoing Laparoscopic Surgery: an Observational Study
Brief Title: The Impact of Anesthesia and Positioning on Cerebral Blood Flow and Pressure in Patients Undergoing Laparoscopic Surgery
Status: Completed | Type: Observational
Sponsor: Xiaguang Duan (Other)
Responsible Party: Sponsor-Investigator, Xiaguang Duan, associate professor (university post), Inner Mongolia Baogang Hospital
Organization: Inner Mongolia Baogang Hospital (Other)
Other Study IDs: 2023-MER-26
Record Dates: First submitted 2024-10-28; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2023-01

CONDITIONS: Laparoscopic Surgery
Keywords: intracranial pressure; laparoscopic; optic nerve sheath diameter; ReverseTrendelenburg position; Trendelenburg position
MeSH Terms: interventions — Pneumoperitoneum, Artificial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- the TREND group (Trendelenburg position): In the Trendelenburg position, the operating table was tilted head down at an angle of 20-25°.
  Interventions: Device: operating position; Device: pneumoperitoneum
- the Reverse Trendelenburg position: In the Reverse Trendelenburg position, the operating table was tilted head up at an angle of 20-25°
  Interventions: Device: operating position; Device: pneumoperitoneum

INTERVENTIONS:
Device: operating position — In the Trendelenburg position, the operating table was tilted head down at an angle of 20-25°. In the Reverse Trendelenburg position, the operating table was tilted head up at an angle of 20-25°.
  Other Names: the Trendelenburg position; the Reverse Trendelenburg position
Device: pneumoperitoneum — Pneumoperitoneum was established with an intra-abdominal pressure of 10-15 mmHg.

SUMMARY:
The aim of this observational study was to understand the effect of ReverseTrendelenburg position, Trendelenburg position on intracranial pressure and carotid blood flow in patients undergoing laparoscopic surgery. The main question it aims to answer is:

Does ReverseTrendelenburg position increase common carotid artery (CCA) flow, optic nerve sheath diameter (ONSD); does Trendelenburg position decrease CCA flow, ONSD.

DETAILED DESCRIPTION:
This study was approved by the Medical Ethics Committee of Inner Mongolia Baogang Hospital, on January 11, 2023 (2023-MER-26)，follow the Declaration of Helsinki. All participants voluntarily agreed to participate and signed informed consent forms. Between February 2023 and December 2023, 76 patients, all classified as ASA I-II adults, were selected at Baogang Hospital, Inner Mongolia. Patients were excluded if they had an allergy to anesthetics used in this study or experienced adverse reactions to analgesics included in the study. Patients were deemed ineligible for clinical evaluation if they refused to sign the consent form or were uncooperative. We excluded patients with a body mass index (BMI) ≥30 kg m-2, uncontrolled hypertension, uncontrolled diabetes, cirrhosis or renal impairment, cardiopulmonary insufficiency, cerebrovascular disease, glaucoma, persistent eye infections, or a history of ophthalmic surgery.

Upon entering the operating room, patients were monitored for pulse oximetry, ECG, BIS, and non-invasive arterial blood pressure. Prior to surgery, patients were administered Penehyclidine Hydrochloride Injection (Lot H20051948, Chengdu List Pharmaceutical Co., Ltd., China) at a dose of 0.01 mg kg-1i.v.. Patients were induced with propofol (1.5-2 mg kg-1i.v.), rocuronium (1-2 mg kg-1i.v.), and fentanyl (1-2μg kg-1i.v.). Anesthesia was maintained with inhaled sevoflurane or desflurane, with inhalation concentrations adjusted according to BIS. Remifentanil (0.05-0.2μg kg-1 min-1i.v.) was continuously infused, with blood pressure and heart rate adjusted to ±20% of baseline values. After induction, patients were mechanically ventilated using the Pressure-Regulated Volume Control (PRVC) mode. Ventilator parameters were set as tidal volume 6-8 ml kg-1, PEEP 0 cmH2O, I ratio of 1:2, respiratory rate 16 breaths per minute (BPM), and FiO2 of 41%. In the Trendelenburg position, the operating table was tilted head down at an angle of 20-25°. In the Reverse Trendelenburg position, the operating table was tilted head up at an angle of 20-25°. Pneumoperitoneum was established with an intra-abdominal pressure of 10-15 mmHg.

Measurements were recorded at five time points: before anesthesia (T1), after intubation (T2), after position change (Trendelenburg or Reverse Trendelenburg position) (T3), after pneumoperitoneum (T4), and at the end of surgery (T5)( Fig 1 b). Parameters measured included mean arterial pressure (MAP; calculated as diastolic pressure + 1/3 pulse pressure), heart rate (HR), Bispectral Index (BIS), PIP, end-tidal carbon dioxide (ETCO2), tidal volume (TV), common carotid artery (CCA) flow, CCA beat volume, CCA diameter, and optic nerve sheath diameter (ONSD). CCA flow, CCA beat volume, CCA diameter, and ONSD were measured using ultrasound by a trained researcher. Ultrasound measurements were performed using the LOGIQ™ E20 device (GE Healthcare, Chicago, Illinois, USA) equipped with a linear 7.5 MHz ultrasound transducer (GE Healthcare, Chicago, Illinois, USA) and a 2.5 MHz ultrasound transducer (GE Healthcare, Chicago, Illinois, USA) to assess optic nerve sheath diameter and common carotid artery blood flow. For each time point, three measurements were taken, and the average value was recorded. Other data were recorded by the anesthesiologist or anesthesia nurse.

In the Postanesthetic Care Unit (PACU), the following parameters were monitored and recorded: length of stay, mean arterial pressure, heart rate, postoperative nausea and vomiting, pain, rescue antiemetics, rescue analgesics, and rescue sulfentanil dose.

ELIGIBILITY:
Inclusion Criteria:

* agreed to participate and signed informed consent forms
* classified as ASA I-II adults

Exclusion Criteria:

* allergy to anesthetics
* refused to sign the consent form or were uncooperative
* a body mass index (BMI) ≥30 kg m-2
* uncontrolled hypertension
* uncontrolled diabetes
* cirrhosis or renal impairment
* cardiopulmonary insufficiency
* persistent eye infections, or a history of ophthalmic surgery

Ages: 29 Years to 62 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Between February 2023 and December 2023, 76 patients, all classified as ASA I-II adults, were selected at Baogang Hospital, Inner Mongolia.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
common carotid artery (CCA) flow | From February 2023 to December 2023
  If it was significantly lower than pre-anesthetic, it was considered that the position and pneumoperitoneum affected the cerebral blood supply.

SECONDARY OUTCOMES:
optic nerve sheath diameter (ONSD) | From February 2023 to December 2023
  If significantly higher than pre-anesthetic, it is thought that the position and pneumoperitoneum have increased intracranial pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangyu Wang, undergraduate, Principal Investigator — Inner Mongolia Baogang Hospital
Locations (1):
- Inner Mongolia Baogang Hospital, Baotou, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: Yes
Recorded parameters were taken at five time points: before anesthesia (T1), after intubation (T2), after positional change (Trendelenburg or Reverse Trendelenburg) (T3), after pneumoperitoneum (T4), and at the end of surgery (T5). Recorded parameters included mean arterial pressure (MAP), heart rate (HR), Bispectral index(BIS), Peak inspiratory pressure (PIP), end-tidal carbon dioxide concentration (ETCO2), Total volume (TV), common carotid artery (CCA) flow, CCA beat volume, CCA diameter, and optic nerve sheath diameter (ONSD).
Supporting Information: Study Protocol, SAP, CSR
Time Frame: January 2025-January 2026